CLINICAL TRIAL: NCT00194571
Title: Helping the Mother With Breast Cancer Support Her Child
Brief Title: Enhancing Connections: Helping the Mother With Breast Cancer Support Her Child
Acronym: EC R01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Frances M. Lewis, Professor, Family and Child Nursing, University of Washington
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 16636-C; 1R01CA078424-01A1 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2008-01

CONDITIONS: Breast Cancer
Keywords: breast cancer,; child functioning,; parenting,; self-efficacy,; psychoeducational intervention; counseling
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Educational counseling intervention — This intervention involves 5 face to face educational counseling sessions with a specially trained patient educator; sessions are fully manualized and complemented by handouts given to the diagnosed parent.

SUMMARY:
This is a 6-state randomized controlled trial (RCT) that uses a behavioral intervention to enhance parenting skills for school age children when a mother is recently diagnosed with early stage breast cancer. Efficacy analyses will include measures of the child's and mother's psychosocial adjustment, including enhanced parenting quality and skills related to the cancer.

DETAILED DESCRIPTION:
This is a Phase 3 randomized clinical trial of recently diagnosed mothers with local or regional breast cancer and their school age child. After baseline measures are taken, mothers are randomized into either intervention and control group. Intervention participants are given 5, 1-hour at home educational counseling sessions by a specially trained nurse. Control participants are mailed an educational booklet whose content focuses on supportive parenting behaviors that are part of the face to face sessions given to the experimental group.

The theoretical framework for the study derives from Bandura's Social Cognitive Theory, a contextual model of parenting, and stress and coping theory. Efficacy is evaluated through standardized valid and reliable questionnaires of psychosocial functioning in the mother (affect, mood, self-efficacy) and psychosocial functioning in the child (cognitive-emotional functioning, including behavioral problems, anxiety, depressed mood, and cancer-related concerns). Primary study hypotheses will be evaluated comparing pre-posttest measures of the intervention compared to controls at post-test and 1-year follow up.

ELIGIBILITY:
Inclusion Criteria:

* Local or regional breast cancer recently diagnosed
* Able to read and write English
* Has one or more school age child(ren) living at home
* Married to a man or in a committed long-term intimate relationship with a male partner

Exclusion Criteria:

* Non-English speaking
* Advanced stage breast cancer
* Not recently diagnosed
* Single mother

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Estimated)
Dates: Start 1999-06; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Increased parenting skills and confidence by diagnosed mothers | 1-year

SECONDARY OUTCOMES:
Decreased anxiety and depressed mood in diagnosed mothers | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Frances M Lewis, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Almulla HA, Lewis FM, Oxford ML. Development and Psychometric Evaluation of the Children's Illness-Related Concerns Scale. Nurs Res. 2023 Sep-Oct 01;72(5):E172-E179. doi: 10.1097/NNR.0000000000000670. PMID 37625187